CLINICAL TRIAL: NCT03757117
Title: Gender-Affirmative Medical Care to Improve HIV Treatment Cascade Among Transgender Women
Brief Title: Gender-Affirmative Transgender Care to Improve the HIV Treatment Cascade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asociación Civil Impacta Salud y Educación, Peru (Other)
Collaborators: The Fenway Institute (Other); Epicentro (Unknown); amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Féminas
Record Dates: First submitted 2018-07-06; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: HIV-1-infection
Keywords: Peru; Health services; Transgender women; Patient navigation; Implementation science; Gender affirming care; HIV prevention; HIV treatment; HIV care cascade

STUDY DESIGN:
Intervention Model Description: Twelve-month, non-randomized, single-arm, pilot cohort study to assess the feasibility, acceptability, and potential effectiveness of integrating routine HIV prevention and treatment services with gender-affirming care supported by transgender woman community peer health navigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Feminizing hormone therapy and peer navigation
  Interventions: Drug: Feminizing hormone therapy; Behavioral: Peer navigation

INTERVENTIONS:
Drug: Feminizing hormone therapy — Estradiol valerate was initiated at 2 mg PO daily and increased to 4 mg after 4 to 12 weeks
  Antiandrogen therapy with spironolactone started at a dose of 50 mg PO daily and increased every 4 weeks to 200 mg daily
Behavioral: Peer navigation — Transgender women community peer navigation

SUMMARY:
Public health strategies are urgently needed to improve HIV disparities among transgender women, highly burdened by the epidemic globally, including holistic approaches that address those health needs prioritized by the community. To address this urgent need, a three-phase implementation science study of an integrated HIV service delivery model that combined HIV prevention and treatment services with gender-affirming primary medical care for transgender women was implemented in Lima, Peru, supported by peer navigation to improve outcomes across the HIV continuum of care: regular HIV testing for HIV-uninfected participants and linkage to preventive services; and engagement in treatment resulting in viral suppression for HIV-infected participants.

DETAILED DESCRIPTION:
A three-phase sequential implementation science study that culturally tailored an informed consent model of transgender care integrating routine HIV prevention and treatment as part of cross-sex hormone therapy supported by peer health navigators for transgender women was implemented in Lima, Peru.

Adult individuals, ages ≥18 years, assigned a male sex at birth, who identified as male-to-female transgender or on the trans-feminine continuum, regardless of initiation or completion of gender enhancement procedures, were eligible to participate. The study target population was transgender women who were unaware of their HIV serostatus or were living with HIV but not engaged in routine HIV care.

Phase 1. Formative research.

Community Engagement and Education. Following principles of Good Participatory Practice to ensure ethical and scientific integrity, based on the specific needs of the target population and to enhance community engagement, a Task Force composed of transgender women community representatives was convened for the study. The Task Force informed the investigators on community issues, advised on study design, supported development of educational programs and campaigns, and facilitated collaborations with the study population. Tailored annual community engagement and education plans were designed in advance of study implementation to include: (1) formative research for stakeholder identification and educational material validation; (2) community awareness activities; and (3) study communication, including development of educational materials, community consultations, and communication of study results.

Mixed-Methods Formative Research. Formative research was conducted among transgender women to assess: (1) experiences accessing HIV prevention services and engagement in HIV primary care, including facilitators and barriers to medical access; (2) attitudes toward a peer navigation system to increase engagement in HIV care; (3) gender-affirmative procedures (experiences with previous and current use of hormone therapy, both personal experiences and community perspectives); (4) assessment of health care needs related to HIV care and gender-affirmation; and (5) attitudes toward having a dedicated facility to receive gender-affirmative care. Formative research also included healthcare professionals (including medical providers and administrators) to assess: (1) knowledge of and experience providing feminization hormone therapy for transgender woman patients; (2) feasibility and acceptability of providing cross-hormone therapy with the existing public health system; (3) acceptability and willingness to provide cross-sex hormone therapy; and (4) perceptions of stigma and discrimination resulting from providing hormone therapy to transgender women. Both transgender women and healthcare professionals were queried about: (1) perceived acceptability of intervention components; and (2) potential barriers to intervention success.

Training. Formative research informed the development of training plans to educate study providers, peer health navigators, and community stakeholders on the hormone therapy intervention. Transgender women community representatives and healthcare providers received medical education training in health care needs, services, and strategies including a gender affirmative approach to transgender medical care, cross-sex hormone therapy, managing HIV infection, and the peer health navigation to improve linkage and retention in care.

Phase 2. Interventional study.

Study Design. Between October 2016 and April 2017, a 12-month, non-randomized, single-arm, pilot cohort study was implemented in Lima, Peru to assess the feasibility, acceptability, and potential effectiveness of integrating routine HIV prevention and treatment services with gender-affirming care (i.e., feminizing hormone therapy) supported by transgender women community peer health navigators. The study was grounded in an implementation science framework, which aimed to test and translate research to promote evidence-based practices for improving health and well-being. Specific design considerations were given to elements that could be replicated by different institutions, including the Ministry of Health, non-governmental organizations and community-based organizations providing HIV care for transgender women, and/or researchers seeking to develop health interventions culturally tailored to the needs of transgender women.

Recruitment. Purposive sampling through peer-recruitment was used to recruit individuals from the target population who were unaware of their HIV serostatus, believed they were HIV-uninfected, or were living with HIV but not engaged in care. Socially well-connected transgender women members and community leaders acted as peer recruiters inviting fellow transgender women to participate in the study. Peer recruiters conducted outreach work by visiting transgender women-specific socialization venues (e.g., commercial sex work areas, beauty parlors, sporting events, community events), where they approached potential participants and referred them to the study site. This recruitment strategy was complemented by social media initiatives to promote study participation.

Screening. Counselors explained the study objectives to potential participants and obtained written informed consent to be screened for participation, HIV and sexually transmitted infection testing, sample storage for further testing, and contact for future studies. Participants who agreed and provided voluntary informed consent underwent a computer-assisted self-interview (CASI) which included questions on demographics, gender identity, sexual orientation and role, sexual risk behavior, previous HIV testing and diagnosis, history of body enhancement procedures and hormone therapy use, life expectations, problems and barriers perceived due to being transgender women, HIV testing history, and prior engagement in care, if HIV positive. Counselors assisted participants in cases of computer unfamiliarity. Physicians obtained a brief medical history and performed a targeted physical examination, including examination of the genitals, anus, lymph nodes, skin, and oropharynx. A peripheral blood sample was obtained for assessment of HIV, syphilis, hepatitis B virus and hepatitis C virus infection, as well as hematology and biochemistry laboratory tests. Participants underwent oropharyngeal and rectal swabbing, and provided a urine sample for the diagnosis of Neisseria gonorrhoeae and Chlamydia trachomatis infection. An anal cytobrush was used to assess the presence of cytological abnormalities induced by human papillomavirus infection. Participants were asked to provide two sputum samples and undergo a chest x-ray to rule out active tuberculosis. Volunteers were convened to return to the site in 2 weeks for the provision of results and enrollment if they were eligible and agreed to participate.

Enrollment. Peer health navigators remained in contact with screened participants and facilitated their return to the research site for enrollment. At the site, a physician assessed eligibility, which included transgender women who resided in Lima and normal hematology and biochemistry laboratory results. Individuals presenting with active tuberculosis, history of pancreatitis, alcohol or drug consumption or other behavioral health condition that in the opinion of the investigator would interfere with the evaluation of the study objectives, severe medical comorbidity, use of immunosuppressive, nephrotoxic or hepatotoxic therapy were excluded. Volunteers received a detailed explanation of the risks and benefits of the medical intervention. Consenting participants underwent a CASI questionnaire, which included questions about personal and social network support for resilience to societal stigma and discrimination, hormone therapy expectations, and housing. Questions about tuberculosis knowledge and attitudes toward its prevention and treatment were also included. A peripheral blood sample was obtained for assessment of baseline fasting glucose and lipids, estradiol and total testosterone levels. For those enrolled without any contraindications, feminization hormone therapy comprised of spironolactone and estradiol valerate was prescribed and dispensed to all participants.

Follow-up. Participants were asked to return to the site for study visits at months 1, 3, 6, 9 and 12, which included follow-up clinical assessment, laboratory testing, and hormone therapy adherence counseling and education following standard protocols. At quarterly visits, participants also received pre- and post-test counseling and sexual risk behavior reduction education, underwent HIV and syphilis testing, and answered a CASI questionnaire on gender identity and body image sexual risk behavior, substance use, attitudes toward HIV testing, personal and social network support, hormone therapy expectations, mental health, adherence to hormone therapy, and involvement in transgender women community building activities. Hormone therapy was dispensed on site on a monthly basis. Peer health navigation facilitated retention in care by outreach work, social media, and phone contact.

Regimen for Feminizing Hormone Therapy. Estradiol valerate was initiated at 2 mg PO daily and increased to 4 mg after 4 to 12 weeks. Antiandrogen therapy with spironolactone started at a dose of 50 mg daily and increased every 4 weeks to 200 mg daily.

Medical Care for HIV Positives and Diagnosed with Sexually Transmitted Infections (STI). Participants diagnosed with HIV infection were referred to standard Peru Ministry of Health protocol care was offered, including initiation of antiretroviral therapy and assessment of baseline and quarterly plasma HIV-1 RNA and cluster of differentiation 4 (CD4+) lymphocyte cell count monitoring. Participants diagnosed with non-HIV STI received international standard treatment and those susceptible to hepatitis B virus were referred for vaccination.

Laboratory Procedures. HIV antibody screening was conducted on whole blood. Positive samples were sent for confirmatory testing to the Peru National Institute of Health laboratory by means of indirect immunofluorescence, unless a previous positive confirmatory result was identified in the Peru NIH database. Plasma HIV-1 RNA and CD4+ lymphocyte cell count assessments were also conducted at the Peru NIH laboratory. Antibodies to Treponema pallidum were detected using a rapid plasma reagin test and confirmed by a T. pallidum particle agglutination assay. Both hepatitis B virus and anti-hepatitis C virus serologies were tested by means of chemiluminescent microparticle immunoassay. N. gonorrhoeae and C. trachomatis infections were diagnosed by a DNA amplification test. Cytological slides were manually colored using standard papanicolaou staining. Sputum testing for tuberculosis used the Ziehl-Neelsen stain. Hematology, biochemistry and hormone tests were assessed automatically. All laboratory test results were provided to participants within a maximum of 14 days, and those with abnormal tests results were referred to clinical care.

Phase 3. Dissemination of intervention and study results.

When intervention 12-month follow-up was near completion, the study team prepared communication plans for disseminating and interpreting study results. Investigators convened the Task Force, Ministry of Health representatives and scientific stakeholders in a community forum to on the implications of the intervention. In this forum, investigators presented a draft version of "Best Practices" for dissemination of integrated transgender women health care services and asked the audience for input that was further incorporated.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as transgender man-to-woman (e.g., "trans", "transgender", "transvestite", or "in the female trans man-woman spectrum)
* 18 years of age or older
* Unaware of HIV serostatus o living with HIV but not engaged in care
* Be willing and able to provide written informed consent to participate, including the understanding of the importance of adhering to the requirements of the study protocol, especially in incorporating prevention, testing and treatment of HIV/STI with feminization hormone therapy with peer-to-peer healthcare navigator support.
* Residence in the city of Lima
* Laboratory values obtained within 21 days prior to their participation in the study:

  * Absolute neutrophil count ≥ 750 cells/mm3
  * Hemoglobin ≥7.0 g/dL
  * Platelet count ≥50,000 cells/mm3
  * Aspartate aminotransferase, alanine aminotransferase, and alkaline phosphatase ≤5 times below the lower limit of normal
  * Serum lipase ≤1.5 times below the lower limit of normal
  * Serum creatinine ≤1.4 times below the lower limit of normal
  * Calculated creatinine clearance (CrCl) ≥50 mL/min according to the Cockcroft-Gault formula

Exclusion Criteria:

* Medical evaluation resulting in a contraindication of the use of hormone therapy
* Measure of non-conformity with his gender inconsistent with the identity of transgender woman
* Allergy or sensitivity or known hypersensitivity to any component of hormones for feminization or their formulations
* Use or active drug or alcohol dependence that in the investigator's opinion, would interfere with adherence to study requirements
* Active tuberculosis
* History of pancreatitis
* Serious medical or psychiatric condition that in the investigator's opinion, would interfere with the ability to adhere to study requirements
* Current treatment with any of the following drugs:

  * Systemic corticosteroids. A short cycle of less than or equal to 21 days of corticosteroids is allowed
  * Systemic chemotherapeutic agents
  * Systemic hepatotoxic or nephrotoxic agents
  * Immunomodulatory treatments
  * Investigational agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals assigned a male sex at birth, who identified as male-to-female transgender or on the trans-feminine continuum (e.g., "trans", "travesti", "transgender", "transsexual"), regardless of initiation or completion of gender enhancement procedures.
Enrollment: 220 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
HIV viral suppression | Twelve months
  Proportion of HIV positive participants who become HIV virally suppressed after 12 months of follow-up
Knowledge of HIV serostatus | Twelve months
  Proportion of HIV negative participants who know their HIV serostatus after 12 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Javier R Lama, MD, MPH, Principal Investigator — Asociación Civil Impacta Salud y Educación; Sari Reisner, ScD, Principal Investigator — The Fenway Institute; Kenneth H Mayer, MD, Principal Investigator — The Fenway Institute
Locations (1):
- Epicentro, Lima, Peru

IPD SHARING:
Plan to Share IPD: Yes
Once all primary and secondary outcomes were assessed, individual participant data study documents would become available upon request and based on investigators´ decision after evaluation
Supporting Information: Study Protocol, ICF
Time Frame: Study protocol and informed consent forms in Spanish are available upon request
Access Criteria: Individual participant data availability will depend on investigators´ decision after evaluation

REFERENCES:
- [Derived] Lama JR, Mayer KH, Perez-Brumer AG, Huerta L, Sanchez H, Clark JL, Sanchez J, Reisner SL. Integration of Gender-Affirming Primary Care and Peer Navigation With HIV Prevention and Treatment Services to Improve the Health of Transgender Women: Protocol for a Prospective Longitudinal Cohort Study. JMIR Res Protoc. 2019 Jun 27;8(6):e14091. doi: 10.2196/14091. PMID 31250829